CLINICAL TRIAL: NCT03071445
Title: Safety and Effectiveness Evaluation of the Minimal Invasive Deformity Correction (MID-C) System in Adolescent Idiopathic Scoliosis (AIS)
Brief Title: Feasibility Study of MID-C for AIS
Acronym: MID-C
Status: Completed | Type: Observational
Sponsor: Apifix (Industry)
Responsible Party: Sponsor
Other Study IDs: AF-01
Record Dates: First submitted 2017-02-26; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a common disorder of unknown etiology in which the vertebrae and discs gradually develop a curvature that is first detected in patients between 11 and 20 years of age. The deformity is 3-dimensional, with a coronal curve measured from radiographs by the Cobb angle .

The Cobb angle measurement of scoliosis represents the sum of the angular wedging of each vertebra and disc between the superior and inferior end vertebrae . Although a small curve is well tolerated and does not require treatment, a large curve can progress to the point that it is cosmetically unacceptable, interferes with chest wall mechanics, and produces cardiac and pulmonary compromises. The natural history of AIS apparently includes 2 stages: the initiation of the curve and its subsequent progression. The factors responsible for the initiation of the curve are unknown, but the subsequent progression of the curve is clearly associated with the adolescent growth spurt . The primary risk factors for progression include age at onset and the magnitude of the curve; young patients with large curves are at the highest risk .

Although numerous treatment methods have been recommended for patients with AIS, the only accepted treatment includes bracing for skeletally immature patients with curves between 25 and 40 degrees and operative correction with spinal fusion for patients with curves greater than 45 degrees. For many teenagers, the cosmetic and social concerns associated with bracing has caused compliance problems with wearing the brace and many patients only wear the brace at home . While operative intervention completely corrects the scoliosis or rib hump, it eliminates segmental spinal motion, and concentrates stresses at the ends of the fusion potentially leading to disc degeneration and back pain.

Despite satisfactory short-term results of operative instrumentation and fusion, a less invasive technique preserving more motion with a smaller scar represents a major improvement. Realizing this goal is contingent on treating curves early, before they progress to an irreversible deformity, and when there is still enough residual growth and remodeling potential.

ApiFix Ltd has developed a novel implant for less invasive treatment of AIS. The MID-C system is designed to correct the deformity step by step along a period of time, giving the skeletal and soft tissues time to accommodate any incremental correction.

The MID-C System inherent benefits are:

* Only two screws are used
* Incision size is much smaller
* Simpler operation with shorter operative time
* Less complications (attributed to the three points above).
* Minimal spinal mobility loss.

All the device components are made of materials well accepted in the orthopedic field and are fully biocompatible (see Investigator Brochure).

The unique concept of the system and the materials used may provide favorable results as follows: Smaller scare, quicker healing period and better spine mobility over the years.

This study is designed to demonstrate that the MID-C System is safe and effective.

DETAILED DESCRIPTION:
The study is designed as an observational study with a 24-month follow-up period. Consecutive patients undergoing treatment of AIS by the MID-C system in daily practice will be included during a 1-year enrollment period.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescence above and inclusive 11 years old
2. Minimum of 35 degrees Cobb angle, confirmed by X-ray. Lenke type 1 or 5
3. Completed at least 6 months of conservative therapy (e.g., P.T., bracing, traction, or others).
4. Reisser sign of 2 to 4
5. Appropriate candidate for posterior surgical approach
6. Subject has Good general health.
7. Subject has no hypersensitivity and allergies to Titanium
8. Subject guardians willing to sign a written informed consent form (ICF).surgeon

Exclusion Criteria:

1. Cobb angle over 55 degrees
2. Other non idiopathic scoliosis.
3. AIS which is not defined as Lenke type 1 or 5
4. Previous spine surgery.
5. Allergy to any component of the device.
6. Active systemic disease, such as AIDS, HIV, or active infection
7. Back or leg pain of unknown etiology
8. Systemic disease that would affect the subject's welfare or overall outcome of the study.
9. Mentally compromised

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study is designed as a prospective, non randomized, open label study with a 24-month follow-up period. Consecutive patients undergoing treatment of AIS by the MID-C system will be included during a 1-years enrollment period.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
No Device related Serious Adverse Event | 2 years
No significant curve progression above or below the implant | 6 months, 1 year, 2 years

SECONDARY OUTCOMES:
Minimum of 50% deformity correction within 6 months | 6 months
Evaluate the correction period using X-ray | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sergiu Straticiuc-ciongradi, MD, Principal Investigator — Spitalul de Copii Sf. Maria Lasi; Peter Than, MD, Principal Investigator — University of Pecs Medical School Hungary; Gheorghe Burnei, MD, PhD, Principal Investigator — Maria Sklodowska Curie, Bucharest
Locations (3):
- University of Pecs, Pécs, Hungary
- Romania (2):
  - Spitalul de Copii Sf. Maria, Iași, Romania
  - Maria Sklodowska Curie, Bucharest

IPD SHARING:
Plan to Share IPD: No